CLINICAL TRIAL: NCT02298452
Title: Structured Post Market Clinical Follow-up (PMCF) to Evaluate the Quality of a New Hearing Aid Product Generation.
Brief Title: Performance of a Hearing Aid Platform Including Different Styles of Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: KEK 2013-0144
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Hearing Loss, Bilateral or Unilateral
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hearing aid (Other): 172 subjects with a mild hearing loss. 140 subjects with a moderate hearing loss. 70 subjects with a severe/ profound hearing loss.
  Interventions: Device: Hearing aid.

INTERVENTIONS:
Device: Hearing aid. — The hearing aid will be fitted to the individual hearing loss of the subject.

SUMMARY:
The reason for this study is to evaluate a new hearing aid product generation replacing the one on the market. The goal is to evaluate the audiological performance, usability as well as features and functions.

DETAILED DESCRIPTION:
This is a controlled, single blinded comparative study which is conducted monocentric at Phonak Headquarters in Staefa. The focus is to compare a new hearing aid product generation with the one on the market as well as with competitor devices regarding the audiological performance, usability as well as features and functions with the aid of 382 mild to profound hearing impaired subjects (18-90 yrs). The subjects, all of them native (Swiss) German speakers, individually conduct a number of laboratory standard tests and home trials (questionnaires) during nine weeks including weekly appointments of 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* all kinds of hearing loss (sensorineural, conductive, combined)
* all kinds of hearing loss (flat, sloping) which are in the fitting range of the hearing aids
* mother tongue (swiss) german

Exclusion Criteria:

Subjects

* with a reduced mobility unable to attend weekly study appointments
* without access to a number of different hearing situations
* with strongly reduced ability to describe auditory impressions and the usage of the hearing aids
* which are uncooperative so that it is not possible to record a valid pure tone audiogram
* with a strongly reduced dexterity
* with psychological problems
* central hearing disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference of speech intelligibility between devices based on Quest platform and Venture platform for different hearing aid styles | 3 years
  For the objective measurements in laboratory situation, both a standard German speech sentence test in noise (SRT in dB) and a standard German monosyllable word test in quiet (speech discrimination in percent) are used to compare the speech intelligibility for both platforms. The results of the Venture platform of both tests should be at least the same or better than with the Quest platform.

SECONDARY OUTCOMES:
Subjective ratings of speech intelligibility during home trials | 3 years
  For the subjective rating of speech intelligibility, questionnaires are used to compare the current platform Quest with the new platform Venture. The subjective impressions are rated by rating scales (e.g. Speech intelligibility in quiet: everything - most - half - little - nothing).
Subjective ratings of sound quality during home trials | 3 years
  For the subjective rating of sound quality, questionnaires are used to compare the current platform Quest with the new platform Venture. The subjective impressions are rated by rating scales (e.g. Sound quality for speech in quiet: good - dull - sharp - thin - echo - scratchy - unclear - noisy).
Subjective ratings of usability during home trials | 3 years
  For the subjective rating of usability, questionnaires are used to compare the current platform Quest with the new platform Venture . The subjective impressions are rated by rating scales (e.g. Rating of the opening and closing of the battery door: very easy - easy - neither - difficult - very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ebbing, B. Sc., Principal Investigator — Phonak AG
Locations (1):
- Phonak AG, Stäfa, Canton of Zurich, Switzerland